CLINICAL TRIAL: NCT01024374
Title: Avaliação da eficácia de um Produto de Uso tópico Contendo Hidrocortisona no Tratamento de Dermatite seborréica na Face.
Brief Title: Evaluation of the Effectiveness of a Product Containing Topical Hydrocortisone in the Treatment of Seborrheic Dermatitis of the Face
Acronym: 13244/2009
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Allergisa Pesquisa Dermato-Cosmetica LTDA (Industry)
Collaborators: Galderma R&D (Industry)
Responsible Party: Douglas - P&D, Galderma
Other Study IDs: All-E-M-13244-01/02-10-09
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2009-12

CONDITIONS: Seborrheic Dermatitis
MeSH Terms: conditions — Dermatitis, Seborrheic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Clinical single-blind randomized comparison with the overall objective of evaluating the clinical efficacy of the products Nutracort lotion and Nutracort cream in the treatment of seborrheic dermatitis on the face.

Will be held clinical and perceived efficacy assessment and instrumental measurements. Each product will be applied at half face for 7 consecutive days and all applications will be monitored in the research site. 60 volunteers will be recruited.

Evaluations will be held at the following times: T0 - before the initial application of the product; T1 - 24 hours after starting treatment, T2 - 48 hours after starting treatment, T3 - 72 hours after initiation of treatment, T4 - 96 hours after the start treatment, T7 - 7 days after initiation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Subjects with seborrheic dermatitis on both sides of the face
* both sexes
* aged 18 to 60 years
* skin types I through IV.

Exclusion Criteria:

* pregnancy / lactation
* skin condition in the area of application of the product
* diabetes
* immune insufficiency
* subjects that are using systemic corticoids
* subjects that are using immunosuppressors
* skin diseases: vitiligo, psoriasis, lupus, atopic dermatitis
* history of reaction to the product category
* other diseases or medications that might interfere directly in the study or endanger the health of the subject

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy subjects with seborrheic dermatitis on both sides of the face, both sexes, aged 18 to 60 years, skin types I through IV.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2010-04